CLINICAL TRIAL: NCT05811104
Title: Accelerated High-dose Sequential Bilateral Theta Burst Stimulation for Treatment Resistant Depression: A Randomized Double-Blind Sham-controlled Pilot Study
Brief Title: Accelerated High-dose Sequential Bilateral Theta Burst Stimulation for Treatment Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Rajamannar Ramasubbu, Professor (Clinical), University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10021798
Record Dates: First submitted 2023-01-05; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: This will be a randomized, sham-controlled, double-blind single centre study using a 1:1 ratio parallel design. We aim to recruit 40 participants (active=20; sham =20) for this pilot study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, clinical assessors and treatment providers will be blinded to treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Experimental): Bilateral real TBS
  Interventions: Device: Sequential bilateral theta burst stimulation
- Sham stimulation (Sham Comparator): Bilateral Sham stimulation
  Interventions: Device: Sequential bilateral theta burst stimulation

INTERVENTIONS:
Device: Sequential bilateral theta burst stimulation — Three sessions of active or sham bilateral TBS will be delivered daily for 10 days in 2 weeks (no session on weekend) with a total of 30 sessions for each patient. Daily low intensity (90% resting motor threshold) bilateral sequential continousTBS ( cTBI) will be applied first on the right DLPFC (1800 pulses) and then intermittent TBS (iTBS)on the left DLPFC (1800 pulses) with an intersession interval of 60 minutes. We will adopt 1800 pulse per session based on the previous studies. Patients will receive a stimulation of 3600 pulses a session, 10,800 pulses a day and 108,000 pulses in total. After the study, sham group will receive active stimulation following the same protocol

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) and Theta burst stimulation (TBS) are approved by the US. Food and Drug administration (FDA) for the treatment of refractory major depression. TBS is more efficient than rTMS as it requires shorter stimulation time.Studies suggest that the efficacy of TBS could be enhanced and expedited by accelerated protocols (more than once daily sessions) with higher doses of stimulation (>600 TBS pulses up to 3600 pulses per session) and shorter duration of treatment (4-10days). The main objective of this study is to determine the clinical efficacy and safety of accelerated high dose bilateral TBS treatment for patients with treatment resistant depression in comparison to sham stimulation using a randomized double blind clinical trial design.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) accounts for the highest global burden of all mental health disorders, and approximately 50% of depressed patients meet criteria for treatment resistant of depression. Stimulation based therapies have recently become a promising alternative for patients with treatment resistant depression. Repetitive transcranial magnetic stimulation (rTMS) of the dorsolateral prefrontal cortex (DLPFC) is approved by the US. Food and Drug administration (FDA) and has been recommended as a viable treatment option for major depression. Recently, a newer form of rTMS called Theta burst stimulation (TBS) is approved by FDA as it has shown comparable clinical efficacy and safety to rTMS in the treatment of depression. TBS is more efficient than rTMS as it requires shorter stimulation time of ≤ 6min compared to 20-40 min required in conventional rTMS protocol and produces equivalent antidepressant responses.

Studies suggest that the efficacy of TBS could be enhanced and expedited by accelerated protocols (more than once daily sessions ranging from 2-10 sessions/day) higher doses of stimulation (>600 TBS pulses up to 3600 pulses per session) with shorter duration of treatment (4-10days). Recently, an accelerated Stanford Neuromodulation Therapy protocol (10 sessions of iTBS a day for 5 days) with high dose stimulation (90,000 pulses in total) was found to be more effective than sham for severe TRD. This protocol yielded robust results with 69.2% response rates compared to 13% in sham during the 4-week outcome period .

The main goal of this project is to determine the clinical efficacy and safety of accelerated high dose bilateral TBS treatment for TRD in comparison to sham stimulation using a randomized double blind clinical trial design. The second objective is to examine the durability of antidepressant effect of this treatment protocol. Our initial open label study of accelerated high dose bilateral TBS demonstrated efficacy in a small cohort of participants with TRD. This proposed study builds on our initial findings whether the antidepressant efficacy of accelerated high dose bilateral TBS would be significantly greater than an identical schedule of sham stimulation. This pilot study will help to examine the feasibility, acceptability, and tolerability of treatment protocol, and estimate the sample size for the next pivotal trial. Hypotheses: Accounting this is a pilot study using small sample size without power size calculations, it is not designed for hypothesis testing. However, it is predicted that the accelerated bilateral TBS would be clinically effective and safe in the treatment of patients with TRD compared to sham stimulation. Additionally, it is anticipated that the antidepressant effects of this treatment may be durable.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDD (DSM-V)
* Adults in the age range of 18 - 65
* Both sex
* HAMD-17 score of ≥20
* TRD - failure to two antidepressant trial Stage II (Thase and Rush classification)

Exclusion Criteria:

* Post traumatic stress disorder,
* Obsessive compulsive disorder,
* Psychosis
* Bipolar disorder,
* substance abuse disorder,
* autistic spectrum disorder,
* active suicidal behavior
* Epilepsy
* Dementia,
* Movement disorders
* severe head injury
* Brain metallic implants, cardiac pacemakers
* Pregnancy .
* Non-response to prior rTMS, Electroconvulsive treatment, Vagal nerve or Deep brain stimulation or a history of psychosurgery.
* Borderline personality disorder,
* Schizotypal, schizoid & paranoid personality disorder
* Current treatment with anticonvulsants or benzodiazepines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | Baseline to week 4 post treatment
  Mean change in Montgomery Asberg Depression Rating Scale (MADRS) scores (0-60) from baseline to week 4 post treatment. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale-17(HDRS-17) | Baseline to week 4 post treatment
  Mean change in Hamilton Depression Rating Scale-17(HDRS-17) scores (0-52) from baseline to week 4 post treatment. Higher scores mean worse outcome
Quick Inventory of Depressive Symptomatology- Self Report (QIDS-SR) | Baseline to week 4 post treatment
  Mean change in Quick Inventory of Depressive Symptomatology- Self Report (QIDS-SR) scores (0-27) from baseline to week 4 post treatment. Higher scores mean worse outcome.
Columbia scale of suicidal behavior (CSS) | Baseline to week 4 post treatment
  Mean change in Columbia scale of suicidal behavior (CSS) scores (2-25) from baseline to week 4 post treatment. Higher scores mean worse outcome.
World Health Organization Quality of Life ( WHOQOL) BREF | Baseline to week 4 post treatment
  Mean change in Quality of Life- ( WHOQOL) BREF - scores ( 0-100) from baseline to week 4 post treatment. Higher scores mean better outcome.
Clinical Global Impression Scale (CGI) | Baseline to week 4 post treatment
  Mean change from Clinical Global Impression Scale (CGI) ( 1-7) baseline to week 4 post treatment. Higher scores mean worse outcome
Categorical outcomes | At 4 week post treatment
  Response (a reduction ≥ 50% in MADRS from the baseline to 4 weekend point) and remission (MADRS score ≤ 10) rates for each group

CONTACTS AND LOCATIONS:
Overall Officials: Rajamannar Ramasubbu, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lisanby SH, Husain MM, Rosenquist PB, Maixner D, Gutierrez R, Krystal A, Gilmer W, Marangell LB, Aaronson S, Daskalakis ZJ, Canterbury R, Richelson E, Sackeim HA, George MS. Daily left prefrontal repetitive transcranial magnetic stimulation in the acute treatment of major depression: clinical predictors of outcome in a multisite, randomized controlled clinical trial. Neuropsychopharmacology. 2009 Jan;34(2):522-34. doi: 10.1038/npp.2008.118. Epub 2008 Aug 13. PMID 18704101
- [Result] Thomas L, Kessler D, Campbell J, Morrison J, Peters TJ, Williams C, Lewis G, Wiles N. Prevalence of treatment-resistant depression in primary care: cross-sectional data. Br J Gen Pract. 2013 Dec;63(617):e852-8. doi: 10.3399/bjgp13X675430. PMID 24351501
- [Result] Levkovitz Y, Isserles M, Padberg F, Lisanby SH, Bystritsky A, Xia G, Tendler A, Daskalakis ZJ, Winston JL, Dannon P, Hafez HM, Reti IM, Morales OG, Schlaepfer TE, Hollander E, Berman JA, Husain MM, Sofer U, Stein A, Adler S, Deutsch L, Deutsch F, Roth Y, George MS, Zangen A. Efficacy and safety of deep transcranial magnetic stimulation for major depression: a prospective multicenter randomized controlled trial. World Psychiatry. 2015 Feb;14(1):64-73. doi: 10.1002/wps.20199. PMID 25655160
- [Result] Blumberger DM, Vila-Rodriguez F, Thorpe KE, Feffer K, Noda Y, Giacobbe P, Knyahnytska Y, Kennedy SH, Lam RW, Daskalakis ZJ, Downar J. Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692. doi: 10.1016/S0140-6736(18)30295-2. Epub 2018 Apr 26. PMID 29726344
- [Result] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062
- [Result] Voigt JD, Leuchter AF, Carpenter LL. Theta burst stimulation for the acute treatment of major depressive disorder: A systematic review and meta-analysis. Transl Psychiatry. 2021 May 28;11(1):330. doi: 10.1038/s41398-021-01441-4. PMID 34050123